CLINICAL TRIAL: NCT00249379
Title: The Use of Acamprosate for Preventing Alcohol Relapse Among Alcohol Dependent Drug Treatment Court Participants
Brief Title: Study of Acamprosate to Prevent Alcohol Relapse in Criminal Justice Supervisees
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Not enough sugjects enrolled before funding ran out
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIAAAWEA-K23-00222-B; K23AA000222 (NIH)
Record Dates: First submitted 2005-11-04; First posted 2005-11-07 (Estimated); Results first posted 2016-05-11 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-04

CONDITIONS: Alcohol Dependence
Keywords: Alcohol dependence; Acamprosate(drug); Drug Court; Probation; Parole; Criminal justice
MeSH Terms: conditions — Alcoholism | interventions — Acamprosate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acamprosate (Experimental): Subjects randomized to receive acamprosate
  Interventions: Drug: Acamprosate
- No medication (No Intervention): No medication intervention (subjects do not receive acamprosate), but do receive Building Social Networks counseling

INTERVENTIONS:
Drug: Acamprosate — Subjects randomized to receive acamprosate 333 mg tablets to be taken 3 times daily to prevent relapse to alcohol dependence
  Other Names: Campral
  Arms: Acamprosate

SUMMARY:
The purpose of this study is to test how tolerable and effective acamprosate is when used to prevent alcohol relapse in criminal justice supervisees (those on probation, parole, or in drug court).

DETAILED DESCRIPTION:
Acamprosate has been an available treatment for alcohol dependence outside the United States and has recently been approved by the U.S. Food and Drug Administration as an effective therapy for alcohol dependence. In the past ten years, drug court programs have been implemented as one possible solution to reduce the burden placed on state and federal correctional systems. These programs are generally focused on non-violent drug dependent offenders and are offered as an alternative to incarceration. However, the use of acamprosate has never been examined for alcohol relapse prevention among a drug court population, or among those on probation or parole.

Comparison: Alcohol-dependent criminal justice supervisees who receive acamprosate, compared to participants who do not receive acamprosate.

ELIGIBILITY:
Inclusion Criteria:

* History of alcohol dependence in the year before entering criminal justice supervision
* Currently under criminal justice supervision (drug court, probation, or parole) in central Virginia

Exclusion Criteria:

* Pregnant or nursing a baby
* Known sensitivity to acamprosate
* Elevated serum creatinine level or other evidence of kidney problems
* Symptoms of severe depression or suicidal ideation
* Non-English speaking such that they cannot provide informed consent
* Cognitive impairment such that they cannot provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2005-06; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael F. Weaver, MD, Principal Investigator — Virginia Commonwealth University Medical Center
Locations (1):
- Virginia Commonwealth University Medical Center, Richmond, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Acamprosate: Criminal justice supervisees given acamprosate 333 mg, 2 tablets orally 3 times daily for alcohol dependence for a 12-week period
- Control: No specific intervention, received standard Drug Court counseling, monitored for outcomes
Period: Overall Study
Arm/Group | Acamprosate | Control
Started | 14 | 12
Completed | 6 | 4
Not Completed | 8 | 8

BASELINE CHARACTERISTICS:
Groups:
- Acamprosate: Criminal justice supervisees given acamprosate for alcohol dependence
- Control: No specific intervention, monitored for outcomes
- Total: Total of all reporting groups
Arm/Group | Acamprosate | Control | Total
Number analyzed (Participants) | 14 | 12 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 12 | 26
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.9 (3) | 37.9 (3) | 37.9 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 10 | 9 | 19
Region of Enrollment [Number; unit: participants]
  United States | 14 | 12 | 26

OUTCOME MEASURES:

1. Primary Outcome: Drinking and Other Drug Use
Description: Number of participants using alcohol and other drugs during 12 weeks
Time Frame: 12 weeks
Population: Only 13 Acamprosate participants were analyzed because one participant was lost to follow-up after being given an initial supply of medication for the study.
  No data were collected for the Control Arm because funding ran out for the study.
Measure: Number; unit: participants
Groups:
- Acamprosate: participants taking study medication
Arm/Group | Acamprosate | Control
Number analyzed (Participants) | 13 | 0
participants | 6 |

2. Primary Outcome: Level of Acceptance
Description: Number of participants taking study medication during 12 weeks
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Acamprosate | Control
Number analyzed (Participants) | 13 | 0
participants | 13 |

3. Secondary Outcome: Retention in Drug Court
Description: Number of participants remaining in drug treatment court program during 12 weeks
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Acamprosate | Control
Number analyzed (Participants) | 13 | 0
participants | 13 |

4. Secondary Outcome: Recidivism Rates
Description: Number of participants returning to jail during 12 weeks
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Acamprosate | Control
Number analyzed (Participants) | 13 | 0
participants | 5 |

ADVERSE EVENTS:
Arm/Group | Acamprosate | Control
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/12
Other Adverse Events (participants affected / at risk) | 0/14 | 0/12

LIMITATIONS AND CAVEATS:
Small numbers of subjects, significant number withdrew or were lost to follow-up

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes